CLINICAL TRIAL: NCT07358663
Title: Assessment of Treatment Outcomes for Esophageal and Gastric Varices Secondary to Portal Hypertension
Brief Title: Treatment Outcomes for Portal Hypertension Esophageal and Gastric Varices
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2025-366
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Esophagogastric Varices; Portal Hypertension
Keywords: endoscopic treatment; portal hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic treatment group: Patients who receive endoscopic treatment
- Non-endoscopic treatment group: Patients who received alternative treatments (excluding endoscopic therapy)

SUMMARY:
This study is a single-center, prospective cohort study based on real-world data. Patients with portal hypertension and esophagogastric varices were enrolled and divided into an endoscopic treatment group and a non-endoscopic treatment group (including patients receiving medical therapy, interventional procedures, or surgical treatment) according to whether they underwent endoscopic intervention. Baseline data, serum metabolites, CT imaging and endoscopic images, liver biopsy pathology, and other multi-omics data were integrated for both groups. Patients were followed up to compare adverse events after variceal treatment, including rebleeding and its causes, hepatic encephalopathy, ascites, subsequent treatments (such as regular endoscopic therapy, NSSB, and TIPS), and survival outcomes. Clinical characteristics of portal hypertension attributed to different etiologies, including hepatitis B, autoimmune liver disease, schistosomiasis, hematological disorders, and chemotherapy-induced liver injury, were compared. The efficacy and safety of endoscopic and interventional treatments for esophagogastric varices were evaluated. Factors influencing rebleeding rates among different treatment groups were analyzed, and reasons for inclusion in different groups were discussed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of portal hypertension with esophagogastric varices.
* Underwent abdominal CT and gastroscopy examinations.

Exclusion Criteria:

* Presence of peptic ulcer, gastric tumor, or other causes of gastrointestinal bleeding confirmed by imaging or gastroscopy.
* CT images of inadequate quality or incomplete medical history data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with portal hypertension and esophagogastric varices between January 2026 and December 2027 were included. Portal hypertension was defined as elevated portal pressure caused by various etiologies, including chronic viral hepatitis, metabolic-associated fatty liver disease, autoimmune liver disease, chemotherapy-induced liver injury, and hematological disorders. The diagnosis of portal hypertension and esophagogastric varices was confirmed by laboratory tests and imaging studies.
Sampling Method: Non-Probability Sample
Enrollment: 1384 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | At 1, 2, 6, and 12 months post-treatment
  Survival status

SECONDARY OUTCOMES:
Adverse events | At 1, 2, 6, and 12 months post-treatment
  Post-treatment adverse events included rebleeding (and its causes), hepatic encephalopathy, and ascites

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Ph.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China